CLINICAL TRIAL: NCT00621725
Title: A Phase I, Open Label Study of the Pharmacokinetics and Safety of Cediranib (RECENTINTM, AZD2171) Following Single and Multiple Oral Doses in Patients With Advanced Solid Tumours With Various Degrees of Hepatic Dysfunction
Brief Title: Phase 1 PK Study of Cediranib in Single and Multiple Doses in Hepatically Impaired Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00032; EUDRACT number 2007-005145-38
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancer; Hepatic Impairment
Keywords: Advanced cancer; metastatic; hepatic impairment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD2171

INTERVENTIONS:
Drug: AZD2171 — Oral dose
  Other Names: Cediranib

SUMMARY:
To determine how patients with advanced cancer and various degrees of hepatic impairment will metabolise Cediranib.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Advanced solid tumour (not prostate cancer) for which no standard therapy exists
* WHO performance status 0-2
* Bilirubin levels within the target range

Exclusion Criteria:

* Unstable brain/meningeal metastases
* Inadequate bone marrow reserve
* Biochemistry/haematology results outside of required ranges
* History of significant GI impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To assess the single dose pharmacokinetics (PK) of Cediranib, in patients with cancer with various degrees of hepatic dysfunction (defined by bilirubin levels). | Single dose PK assessed on Day 1 of dosing

SECONDARY OUTCOMES:
Safety/tolerability of Cediranib (single and multiple dose PK) | assessed from randomisation to data cut-off (15th July 2010)
  Single and multiple dose PK assessed on Day 1 of the single dosing period and Day 21 of the multiple dosing period, respectively (minimum 7 day washout following single dosing)

CONTACTS AND LOCATIONS:
Overall Officials: CML van Herpen, MD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Research Site, København Ø, Denmark
- Netherlands (2):
  - Research Site, Nijmegen
  - Research Site, Rotterdam

REFERENCES:
- [Derived] van Herpen CM, Lassen U, Desar IM, Brown KH, Marotti M, de Jonge MJ. Pharmacokinetics and tolerability of cediranib, a potent VEGF signalling inhibitor, in cancer patients with hepatic impairment. Anticancer Drugs. 2013 Feb;24(2):204-11. doi: 10.1097/CAD.0b013e32835bd1d2. PMID 23197081
- See also: CSR-D8480C00032.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=629&filename=CSR-D8480C00032.pdf